CLINICAL TRIAL: NCT04205331
Title: Validity Of Ultrasound As Regards Correlation To Cormack-Lehane Grading In Obese Patients: A Cross Sectional Observational Study
Brief Title: Validity Of Ultrasound As Regards Correlation To Cormack-Lehane Grading In Obese Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed Abdelrahman Mohamed El-Tawansy, Principal Investigator, Zagazig University
Other Study IDs: 5162-23-1-2019
Record Dates: First submitted 2019-12-14; First posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Difficult Airway Intubation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- obese patients: compare between ultrasonography and conventional clinical methods of airway assessment prior to induction of anesthesia correlating it to the Cormack-Lehane scoring system after induction of anesthesia in obese patients
  Interventions: Device: Assessing validity of ultrasound as regards correlation to Cormack-Lehane grading in obese patients

INTERVENTIONS:
Device: Assessing validity of ultrasound as regards correlation to Cormack-Lehane grading in obese patients — Assessing validity of ultrasound as regards correlation to Cormack-Lehane grading in obese patients

SUMMARY:
Since the introduction of real-time ultrasound (US) capabilities, ultrasound technology has been adopted and incorporated into daily practice by many medical and surgical specialties. Using US to help assess the difficult airway constitutes just yet another valuable application of this versatile technology . Since many anesthesia providers had already acquired proficiency in US techniques in US guided vascular access and regional nerve blocks, using US to evaluate the airway could be learned and mastered without too much difficulty. Ultrasound of the upper airway may prove to become a useful adjunct to conventional clinical assessment tools, as it has been successful in visualizing the relevant anatomy and critical structures of the airway..

DETAILED DESCRIPTION:
The study is cross sectional observational study in which obese patients will be assessed using conventional clinical methods of airway assessment and by using US for the same patient before induction of anesthesia then correlated to the Cormack-Lehane finding after induction of anesthesia..

ELIGIBILITY:
Inclusion Criteria:

* Age of the patient : (21-60) years old.
* Sex : male & female.
* Physical Status : The American Society of Anesthesiologists (ASA) II-III patients.
* Body mass index : 30 to more than 30 kg / m² .
* Operations: Laparoscopic surgeries,bariatric surgeries and any operation that requires general anesthesia with endotracheal tube placement .

Exclusion Criteria:

Patient refusal.

* Deformity of the airway anatomy [by masses or tumors].
* Patients with thyroid swellings 'Goitre'.
* Pathology of the airway [edema,burn and arthritis].

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will be conducted at Zagazig University Hospitals.The study is cross sectional observational study in which obese patients will be assessed using conventional clinical methods of airway assessment and by using US for the same patient before induction of anesthesia then correlated to the Cormack-Lehane finding after induction of anesthesia.
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2019-12-14 (Actual); Primary Completion 2020-09-20 (Estimated); Study Completion 2020-10-20 (Estimated)

PRIMARY OUTCOMES:
The ratio of the depth of the pre-epiglottic space (Pre-E) to the distance from the epiglottis to the mid-point of the distance between the vocal cords (E-VC). | through study completion, an average of 1 year
  If It is [0-1] ,this suspects Cormack-Lehane Grade 1.If it is [1-2],this suspects Cormack-Lehane Grade 2.If it is [2-3],this suspects Cormack-Lehane Grade 3
The anterior neck soft tissue thickness at the level of the vocal cords (ANS-VC) | through study completion, an average of 1 year
  ANS-VC >0.23 cm had a sensitivity of 85.7% in predicting a Cormack-Lehan Grade 3 or 4

SECONDARY OUTCOMES:
The anterior neck soft tissue thickness at the level of the hyoid bone (ANS-Hyoid) | through study completion, an average of 1 year
  If it is 1.69 cm [1.19 cm to 2.19 cm],this suspects difficult laryngoscopy.If it is 1.37cm [1.27 cm to 1.46 cm], this suspects easy laryngoscopy
The hyomental distance of the patient in neutral position of the neck and in fully extended neck calculating the ratio between both of them | through study completion, an average of 1 year
  If The mean hyomental distance ratios is (1.02 ± 0.01) ,this suspects difficult intubation.If it is (1.14 ± 0.02) ,this suspects easy intubation
Tongue volume will be derived from multiplication of the midsagittal cross-sectional area of the tongue by its width obtained from transverse sonograms | through study completion, an average of 1 year
  Large tongue volume suspects difficult laryngoscopy
Modified Mallampati classification | through study completion, an average of 1 year
  Class I is visualization of the hard palate, soft palate, fauces, uvula, and pillars.
  Class II is visualization of the hard palate, soft palate, fauces, and base of uvula.
  Class III is visualization of the hard palate and soft palate. Class IV is visualization of only the hard palate
Interincisor gap | through study completion, an average of 1 year
  If it is less than 5 cm (approximately three finger breadths) with limited forward protrusion of the mandible ,this is associated with increased risk of difficult laryngoscopy
Thyromental distance | through study completion, an average of 1 year
  If < 6cm ,this predicts difficult laryngoscopy
Sternomental distance | through study completion, an average of 1 year
  If < 12.5 cm ,this predicts difficult laryngoscopy
Neck Extension and Flexion | through study completion, an average of 1 year
  inability to extend or flex the neck suspects difficult laryngoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El-Tawansy, M.Sc., Principal Investigator — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Protocol and Results will be shared with other researchers.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication
Access Criteria: anesthesiologists who are interested in airway management